CLINICAL TRIAL: NCT04632537
Title: Novel Use of an Existing Vaccine (BCG) Alliance: The NUEVA Trial
Brief Title: BCG Vaccination to Prevent COVID-19
Acronym: NUEVA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to funding - project never enrolled
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Defense Health Agency (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: USUHS.2020-062
Record Dates: First submitted 2020-11-04; First posted 2020-11-17 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: COVID-19; BCG; vaccine; clinical trial
MeSH Terms: conditions — COVID-19 | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TICE BCG (for intravesical use, Merck) BCG LIVE (Active Comparator): Participants randomized to the BCG arm will receive Tice® BCG (for intravesical use) BCG LIVE is a live freeze-dried vaccine made from an attenuated strain of Mycobacterium bovis. The freeze-dried vaccine will be delivered in vials, each containing 1 to 8 x108 colony forming units (CFU). Tice® BCG (for intravesical use) BCG LIVE will be reconstituted in ~5 mL of preservative-free saline, as needed for yielding 2- x107 CFU/ mL. [34] Administration of 0.1 mL will contain 2x106 CFU, which accounts for approximately 0.1 mg of the attenuated Mycobacterium bovis. Administration of 0.1 mL of diluted vaccine will be given per dose, intradermally. A sterile tuberculin 1mL syringe and sterile fine short needle (25 or 26 gauge with 3/8-3/4 length), will be used for each injection. The injection should be made slowly after inserting the needle ~2 mm into the superficial layer of the dermis of the upper arm (usually deltoid area), to make a symmetrical superficial bleb.
  Interventions: Drug: Tice® BCG (for intravesical use) BCG LIVE strain of the BCG (Merck) vaccine
- placebo vaccine (Placebo Comparator): Placebo will be administered in an intradermal route in the same location as the BCG vaccines: upper arm. Placebo will comprise 0.1 mL of the diluent (preservative-free saline) to ensure the same quantity and same color as the resuspended BCG vaccine, rendering the two indistinguishable.
  Interventions: Drug: Preservative-free saline

INTERVENTIONS:
Drug: Tice® BCG (for intravesical use) BCG LIVE strain of the BCG (Merck) vaccine — Tice® BCG (for intravesical use) BCG LIVE strain of the BCG (Merck) vaccine will be diluted in preservative-free saline and given intradermally (0.1mL) in the deltoid area.
  Arms: TICE BCG (for intravesical use, Merck) BCG LIVE
Drug: Preservative-free saline — Placebo will be administered in an intradermal route in the same location as the BCG vaccines: upper arm. Placebo will comprise 0.1 mL of the diluent (preservative-free saline) to ensure the same quantity and same color as the resuspended BCG vaccine, rendering the two indistinguishable.
  Arms: placebo vaccine

SUMMARY:
The current COVID-19 epidemic threatens to overwhelm the capacity of many countries to meet their populations' health care needs. Although several vaccines specific for SARS-CoV-2 have been or are being developed, these require testing in animal and human safety studies and they are unlikely to be available during the expected peak periods of the growing epidemic. Two groups at especially high risk of infection and disease are front line health care workers working directly with COVID-19 patients and elderly residents of group homes or facilities that provide skilled nursing care to this frail population. Interim measures to protect these groups while we await a high efficacy vaccine are desperately needed.

Based on the capacity of BCG to (1) reduce the incidence of respiratory tract infections in children and adults; (2) exert antiviral effects in experimental models; and (3) reduce viremia in an experimental human model of viral infection, we hypothesize that BCG vaccination may induce (partial) protection against susceptibility to and/or severity of SARS-CoV-2 infection.

This study will evaluate the efficacy of BCG to reduce risk of infection by SARS-CoV-2 and mitigate COVID-19 disease severity in at risk health care providers.

A phase III randomized controlled trial provides the highest validity to answer this research question. Given the immediate threat of the SARS-CoV-2 epidemic the trial has been designed as a pragmatic study with a highly feasible primary endpoint, which can be continuously measured. This allows for the most rapid identification of a beneficial outcome that would allow other at-risk individuals, including the control population, to also benefit from the intervention if and as soon as it has demonstrated efficacy and safety.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, double-blind, randomized placebo-controlled trial to assess the efficacy of intradermal TICE BCG (for intravesical use, Merck) BCG LIVE or placebo vaccine, in reducing the incidence of infection of SARS-CoV2 and severity of COVID-19 disease. This study proposes to examine BCG-induced nonspecific trained immunity to provide protection from SARS-CoV2 among health care workers who are likely to care for patients with COVID-19 illness, 18-64 years of age.

Up to 670 individuals will be screened to enroll 550 participants with a planned 50 person enrollment at USU site, 300 persons at Darnall Medical Center (CRDMC) and 200 persons at Brooke Army Medical Center (BAMC), resulting in 275 receiving BCG vaccine and 275 receiving placebo. To account for attrition prior to vaccination we will enroll up to 70 at USU, up to 350 at CRDMC and up to 250 at BAMC.

There are three phases in which research procedures will be completed: (1) initial screening for eligibility, consent, baseline testing; (2) enrollment, randomization, if pertains- prior to vaccination research blood draw for peripheral blood mononuclear cells (PBMC), and immunization with study vaccine (BCG or placebo); and (3) follow-up screening and testing.

Participants will be followed to assess whether infection with SARS-CoV-2 occurs:

Participants will complete intermittent surveys via an electronic system every 2 weeks to assess the presence of any flu-like symptom. Any positive response on the survey will trigger a nasopharyngeal swab to be collected to test for COVID-19 via rt-PCR.

All participants, regardless of survey responses, will have serology (4mL SST tube) for COVID-19 tested at monthly intervals during the 6 month follow-up period or until a positive test result occurs.

If a participant completes the follow-up period and does not test positive for COVID disease, study participation is complete.

If a participant does test positive for COVID-19 disease at any point during follow-up, disease status will be ascertained for up to two months from the time of positive test or until an outcome is available through one of the following mechanisms:

(1) an electronic survey if not admitted to the hospital, including questions about the number of days ill, daily fever, and other symptoms; or (2) if admitted to the hospital, ordinal outcomes for disease severity will be extracted from the hospital's medical records system for the 2 month period of highest acuity. Participants will have a final study visit after hospitalization when cleared for outpatient follow up.

During the first 6 weeks of follow-up post vaccination, all participants will be asked about any adverse events; thereafter, participants will report vaccine-related and solicited adverse events (AE), as well as unsolicited AEs through the electronic survey.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, physician assistants, nurse practitioners, nurses, medics, respiratory therapists and other HCWs who are likely to care for patients with COVID-19 illness
* Eligible for care in DoD facilities (DEERS eligible)*
* 18-64 years old
* Willingness to permit review of medical records
* Women of childbearing potential must be willing to use an effective form of birth control for 30 days post vaccination

Exclusion Criteria:

* Previously (medical history) or currently infected or ill with COVID-19
* Previous TB disease
* Fever (>38 C) within the past 24 hours
* Currently pregnant or breastfeeding or planning on becoming pregnant within 30 days of enrollment
* Current serious underlying medical conditions including: diabetes mellitus, chronic kidney disease, or any other immunocompromising condition:

  * Known infection by Human Immunodeficiency Virus (HIV)
  * History of solid organ or bone marrow transplantation
  * Currently under chemotherapy
  * Currently on any anti-cytokine therapy
  * History of immunodeficiency (including history of anti B cell therapy)
  * Currently taking immunosuppressive drugs
  * Treatment with oral or intravenous steroids, defined as daily doses of 10mg prednisone or equivalent for longer than 3 months
* Active solid or non-solid malignancy or lymphoma within the past two years
* Suspicion of active viral or bacterial infection
* Living with someone HIV+, who is immunocompromised, or is taking an immunosuppressive drug
* Known allergy to (components of) the BCG vaccine or a serious reaction to prior BCG administration
* Plan to terminate their employment at the participating health care facility or change duty stations within the next three months
* Not in possession of a smartphone
* Current participation in a COVID-19 interventional trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic rt-PCR-confirmed SARS-CoV-2 infection | 6 months
  The primary outcome measure is the development of symptomatic COVID 19 infections. We will use the Cox proportional-hazards model to calculate hazard ratios for the development of COVID-19. This will be reported as the incidence of rt-PCR-confirmed symptomatic SARS-CoV-2 infection following BCG vaccination compared to that following placebo, starting from 3 days post-vaccination through 6 months.

SECONDARY OUTCOMES:
incidence of Serology-confirmed infection with SARS-CoV-2 | 6 months
  The secondary outcome measure is the development of Serology-confirmed infection with SARS-CoV-2. We will use the Cox proportional-hazards model to calculate hazard ratios for the development of COVID-19. This will be reported as the incidence of serology-confirmed SARS-CoV-2 following BCG vaccination compared to that following placebo, starting from 3 days post vaccination through 6 months.
severity of COVID-19 disease | 6 months
  In individuals who test positive for COVID-19, the proportion with severe disease following BCG vaccination compared to placebo, as defined by the following necessary care levels: non- hospital care; patient hospitalized but no oxygen required; hospitalized and oxygen required; patient treated in intensive care and/or on mechanical ventilation; patient died.Additional WHO severity indicators of severe pneumonia, respiratory failure, sepsis, septic shock will also be included.
symptomatic respiratory infection | 6 months
  Incidence of self-reported symptomatic respiratory infections following BCG vaccination compared to that following placebo, starting from 3 days post-vaccination through 6 months.
effect of prior adult immunization with other vaccines associated with trained immunity | 6 months
  rates of 1) all cause respiratory infection 2) symptomatic COVID- 19, 3) serology-confirmed SARS-CoV-2 infection in health care workers.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Livezey, MD, Principal Investigator — Uniformed Services University of the Health Sciences; Naomi E Aronson, Study Chair — Uniformed Services University of the Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Coronavirus disease 2019 (COVID-19): Situation Report - 23. COVID-19 Situational Reports (2020). Accessed on April 1, 2020 at: https://www.who.int/docs/default- source/coronaviruse/situation-reports/20200212-sitrep-23-nCoV.pdf?sfvrsn=41e9fb78_4
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chang D, Xu H, Rebaza A, Sharma L, Dela Cruz CS. Protecting health-care workers from subclinical coronavirus infection. Lancet Respir Med. 2020 Mar;8(3):e13. doi: 10.1016/S2213-2600(20)30066-7. Epub 2020 Feb 13. No abstract available. PMID 32061333
- [Background] Zhang J, Zhou L, Yang Y, Peng W, Wang W, Chen X. Therapeutic and triage strategies for 2019 novel coronavirus disease in fever clinics. Lancet Respir Med. 2020 Mar;8(3):e11-e12. doi: 10.1016/S2213-2600(20)30071-0. Epub 2020 Feb 13. No abstract available. PMID 32061335
- [Background] Chou R, Dana T, Buckley DI, Selph S, Fu R, Totten AM. Epidemiology of and Risk Factors for Coronavirus Infection in Health Care Workers: A Living Rapid Review. Ann Intern Med. 2020 Jul 21;173(2):120-136. doi: 10.7326/M20-1632. Epub 2020 May 5. PMID 32369541
- [Background] Rivett L, Sridhar S, Sparkes D, Routledge M, Jones NK, Forrest S, Young J, Pereira-Dias J, Hamilton WL, Ferris M, Torok ME, Meredith L; CITIID-NIHR COVID-19 BioResource Collaboration; Curran MD, Fuller S, Chaudhry A, Shaw A, Samworth RJ, Bradley JR, Dougan G, Smith KG, Lehner PJ, Matheson NJ, Wright G, Goodfellow IG, Baker S, Weekes MP. Screening of healthcare workers for SARS-CoV-2 highlights the role of asymptomatic carriage in COVID-19 transmission. Elife. 2020 May 11;9:e58728. doi: 10.7554/eLife.58728. PMID 32392129
- [Background] CDC COVID-19 Response Team. Characteristics of Health Care Personnel with COVID-19 - United States, February 12-April 9, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 17;69(15):477-481. doi: 10.15585/mmwr.mm6915e6. PMID 32298247
- [Background] Nguyen LH, Drew DA, Graham MS, Joshi AD, Guo CG, Ma W, Mehta RS, Warner ET, Sikavi DR, Lo CH, Kwon S, Song M, Mucci LA, Stampfer MJ, Willett WC, Eliassen AH, Hart JE, Chavarro JE, Rich-Edwards JW, Davies R, Capdevila J, Lee KA, Lochlainn MN, Varsavsky T, Sudre CH, Cardoso MJ, Wolf J, Spector TD, Ourselin S, Steves CJ, Chan AT; COronavirus Pandemic Epidemiology Consortium. Risk of COVID-19 among front-line health-care workers and the general community: a prospective cohort study. Lancet Public Health. 2020 Sep;5(9):e475-e483. doi: 10.1016/S2468-2667(20)30164-X. Epub 2020 Jul 31. PMID 32745512
- [Background] Wang X, Ferro EG, Zhou G, Hashimoto D, Bhatt DL. Association Between Universal Masking in a Health Care System and SARS-CoV-2 Positivity Among Health Care Workers. JAMA. 2020 Aug 18;324(7):703-704. doi: 10.1001/jama.2020.12897. PMID 32663246
- [Background] Ritz N, Hanekom WA, Robins-Browne R, Britton WJ, Curtis N. Influence of BCG vaccine strain on the immune response and protection against tuberculosis. FEMS Microbiol Rev. 2008 Aug;32(5):821-41. doi: 10.1111/j.1574-6976.2008.00118.x. Epub 2008 Jul 9. PMID 18616602
- [Background] Abubakar I, Pimpin L, Ariti C, Beynon R, Mangtani P, Sterne JA, Fine PE, Smith PG, Lipman M, Elliman D, Watson JM, Drumright LN, Whiting PF, Vynnycky E, Rodrigues LC. Systematic review and meta-analysis of the current evidence on the duration of protection by bacillus Calmette-Guerin vaccination against tuberculosis. Health Technol Assess. 2013 Sep;17(37):1-372, v-vi. doi: 10.3310/hta17370. PMID 24021245
- [Background] Walk J, de Bree LCJ, Graumans W, Stoter R, van Gemert GJ, van de Vegte-Bolmer M, Teelen K, Hermsen CC, Arts RJW, Behet MC, Keramati F, Moorlag SJCFM, Yang ASP, van Crevel R, Aaby P, de Mast Q, van der Ven AJAM, Stabell Benn C, Netea MG, Sauerwein RW. Outcomes of controlled human malaria infection after BCG vaccination. Nat Commun. 2019 Feb 20;10(1):874. doi: 10.1038/s41467-019-08659-3. PMID 30787276
- [Background] Koeken VACM, Verrall AJ, Netea MG, Hill PC, van Crevel R. Trained innate immunity and resistance to Mycobacterium tuberculosis infection. Clin Microbiol Infect. 2019 Dec;25(12):1468-1472. doi: 10.1016/j.cmi.2019.02.015. Epub 2019 Feb 23. PMID 30807849
- [Background] Suliman S, Geldenhuys H, Johnson JL, Hughes JE, Smit E, Murphy M, Toefy A, Lerumo L, Hopley C, Pienaar B, Chheng P, Nemes E, Hoft DF, Hanekom WA, Boom WH, Hatherill M, Scriba TJ. Bacillus Calmette-Guerin (BCG) Revaccination of Adults with Latent Mycobacterium tuberculosis Infection Induces Long-Lived BCG-Reactive NK Cell Responses. J Immunol. 2016 Aug 15;197(4):1100-1110. doi: 10.4049/jimmunol.1501996. Epub 2016 Jul 13. PMID 27412415
- [Background] Nemes E, Geldenhuys H, Rozot V, Rutkowski KT, Ratangee F, Bilek N, Mabwe S, Makhethe L, Erasmus M, Toefy A, Mulenga H, Hanekom WA, Self SG, Bekker LG, Ryall R, Gurunathan S, DiazGranados CA, Andersen P, Kromann I, Evans T, Ellis RD, Landry B, Hokey DA, Hopkins R, Ginsberg AM, Scriba TJ, Hatherill M; C-040-404 Study Team. Prevention of M. tuberculosis Infection with H4:IC31 Vaccine or BCG Revaccination. N Engl J Med. 2018 Jul 12;379(2):138-149. doi: 10.1056/NEJMoa1714021. PMID 29996082
- [Background] World Health Organization. Clinical Management of Severe acute respiratory infection when COVID-19 is suspected. (2020). Accessed on April 1, 2020 at: https://apps.who.int/iris/bitstream/handle /10665/331446/WHO-2019-nCoV-clinical-2020.4- eng.pdf.
- [Background] O'Neill LAJ, Netea MG. BCG-induced trained immunity: can it offer protection against COVID-19? Nat Rev Immunol. 2020 Jun;20(6):335-337. doi: 10.1038/s41577-020-0337-y. PMID 32393823
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Joosten LA, Ifrim DC, Saeed S, Jacobs C, van Loenhout J, de Jong D, Stunnenberg HG, Xavier RJ, van der Meer JW, van Crevel R, Netea MG. Bacille Calmette-Guerin induces NOD2-dependent nonspecific protection from reinfection via epigenetic reprogramming of monocytes. Proc Natl Acad Sci U S A. 2012 Oct 23;109(43):17537-42. doi: 10.1073/pnas.1202870109. Epub 2012 Sep 17. PMID 22988082
- [Background] Spencer JC, Ganguly R, Waldman RH. Nonspecific protection of mice against influenza virus infection by local or systemic immunization with Bacille Calmette-Guerin. J Infect Dis. 1977 Aug;136(2):171-5. doi: 10.1093/infdis/136.2.171. PMID 894076
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Netea MG, Giamarellos-Bourboulis EJ, Dominguez-Andres J, Curtis N, van Crevel R, van de Veerdonk FL, Bonten M. Trained Immunity: a Tool for Reducing Susceptibility to and the Severity of SARS-CoV-2 Infection. Cell. 2020 May 28;181(5):969-977. doi: 10.1016/j.cell.2020.04.042. Epub 2020 May 4. PMID 32437659
- [Background] Arts RJW, Moorlag SJCFM, Novakovic B, Li Y, Wang SY, Oosting M, Kumar V, Xavier RJ, Wijmenga C, Joosten LAB, Reusken CBEM, Benn CS, Aaby P, Koopmans MP, Stunnenberg HG, van Crevel R, Netea MG. BCG Vaccination Protects against Experimental Viral Infection in Humans through the Induction of Cytokines Associated with Trained Immunity. Cell Host Microbe. 2018 Jan 10;23(1):89-100.e5. doi: 10.1016/j.chom.2017.12.010. PMID 29324233
- [Background] Netea MG, van Crevel R. BCG-induced protection: effects on innate immune memory. Semin Immunol. 2014 Dec;26(6):512-7. doi: 10.1016/j.smim.2014.09.006. Epub 2014 Oct 23. PMID 25444548
- [Background] Kleinnijenhuis J, van Crevel R, Netea MG. Trained immunity: consequences for the heterologous effects of BCG vaccination. Trans R Soc Trop Med Hyg. 2015 Jan;109(1):29-35. doi: 10.1093/trstmh/tru168. PMID 25573107
- [Background] Higgins JP, Soares-Weiser K, Lopez-Lopez JA, Kakourou A, Chaplin K, Christensen H, Martin NK, Sterne JA, Reingold AL. Association of BCG, DTP, and measles containing vaccines with childhood mortality: systematic review. BMJ. 2016 Oct 13;355:i5170. doi: 10.1136/bmj.i5170. PMID 27737834
- [Background] Wardhana, Datau EA, Sultana A, Mandang VV, Jim E. The efficacy of Bacillus Calmette-Guerin vaccinations for the prevention of acute upper respiratory tract infection in the elderly. Acta Med Indones. 2011 Jul;43(3):185-90. PMID 21979284
- [Background] Han RF, Pan JG. Can intravesical bacillus Calmette-Guerin reduce recurrence in patients with superficial bladder cancer? A meta-analysis of randomized trials. Urology. 2006 Jun;67(6):1216-23. doi: 10.1016/j.urology.2005.12.014. PMID 16765182
- [Background] Leentjens J, Kox M, Stokman R, Gerretsen J, Diavatopoulos DA, van Crevel R, Rimmelzwaan GF, Pickkers P, Netea MG. BCG Vaccination Enhances the Immunogenicity of Subsequent Influenza Vaccination in Healthy Volunteers: A Randomized, Placebo-Controlled Pilot Study. J Infect Dis. 2015 Dec 15;212(12):1930-8. doi: 10.1093/infdis/jiv332. Epub 2015 Jun 12. PMID 26071565
- [Background] World Health Organization. Expert committee on biological standardization: Recommendations to assure the quality, safety and efficacy of BCG vaccines. (2011). Accessed on April 1, 2020 at: https://www.who.int/biologicals/BCG_DB_HK_23_April_2012.pdf
- [Background] Hatherill M, Geldenhuys H, Pienaar B, Suliman S, Chheng P, Debanne SM, Hoft DF, Boom WH, Hanekom WA, Johnson JL. Safety and reactogenicity of BCG revaccination with isoniazid pretreatment in TST positive adults. Vaccine. 2014 Jun 30;32(31):3982-8. doi: 10.1016/j.vaccine.2014.04.084. Epub 2014 May 9. PMID 24814553
- [Background] McKee AS, Munks MW, Marrack P. How do adjuvants work? Important considerations for new generation adjuvants. Immunity. 2007 Nov;27(5):687-90. doi: 10.1016/j.immuni.2007.11.003. PMID 18031690
- [Background] Mangtani P, Abubakar I, Ariti C, Beynon R, Pimpin L, Fine PE, Rodrigues LC, Smith PG, Lipman M, Whiting PF, Sterne JA. Protection by BCG vaccine against tuberculosis: a systematic review of randomized controlled trials. Clin Infect Dis. 2014 Feb;58(4):470-80. doi: 10.1093/cid/cit790. Epub 2013 Dec 13. PMID 24336911
- [Background] Kemp EB, Belshe RB, Hoft DF. Immune responses stimulated by percutaneous and intradermal bacille Calmette-Guerin. J Infect Dis. 1996 Jul;174(1):113-9. doi: 10.1093/infdis/174.1.113. PMID 8655980
- [Background] Pizzi M, Albertoni L, Stefanizzi L, Mescoli C, Rugge M. Gastrointestinal Crohn-like disease following BCG therapy. Int J Colorectal Dis. 2015 Dec;30(12):1745-6. doi: 10.1007/s00384-015-2157-2. Epub 2015 Feb 18. No abstract available. PMID 25690704
- [Background] Queiro R, Ballina J, Weruaga A, Fernandez JA, Riestra JL, Torre JC, Rodriguez A. Psoriatic arthropathy after BCG immunotherapy for bladder carcinoma. Br J Rheumatol. 1995 Nov;34(11):1097. doi: 10.1093/rheumatology/34.11.1097. No abstract available. PMID 8542217
- [Background] Dudelzak J, Curtis AR, Sheehan DJ, Lesher JL Jr. New-onset psoriasis and psoriatic arthritis in a patient treated with Bacillus Calmette-Guerin (BCG) immunotherapy. J Drugs Dermatol. 2008 Jul;7(7):684. No abstract available. PMID 18664162
- [Background] Randomised controlled trial of single BCG, repeated BCG, or combined BCG and killed Mycobacterium leprae vaccine for prevention of leprosy and tuberculosis in Malawi. Karonga Prevention Trial Group. Lancet. 1996 Jul 6;348(9019):17-24. PMID 8691924
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Chen Y, Li L. SARS-CoV-2: virus dynamics and host response. Lancet Infect Dis. 2020 May;20(5):515-516. doi: 10.1016/S1473-3099(20)30235-8. Epub 2020 Mar 23. No abstract available. PMID 32213336
- [Background] Hoft DF, Leonardi C, Milligan T, Nahass GT, Kemp B, Cook S, Tennant J, Carey M. Clinical reactogenicity of intradermal bacille Calmette-Guerin vaccination. Clin Infect Dis. 1999 Apr;28(4):785-90. doi: 10.1086/515201. PMID 10825039
- [Background] Giamarellos-Bourboulis EJ, Tsilika M, Moorlag S, Antonakos N, Kotsaki A, Dominguez-Andres J, Kyriazopoulou E, Gkavogianni T, Adami ME, Damoraki G, Koufargyris P, Karageorgos A, Bolanou A, Koenen H, van Crevel R, Droggiti DI, Renieris G, Papadopoulos A, Netea MG. Activate: Randomized Clinical Trial of BCG Vaccination against Infection in the Elderly. Cell. 2020 Oct 15;183(2):315-323.e9. doi: 10.1016/j.cell.2020.08.051. Epub 2020 Sep 1. PMID 32941801